CLINICAL TRIAL: NCT04351100
Title: Efficacy of Diacerein on Ocular Surface Disease in Degenerative Arthritis Patients
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Ngamjit Kasetsuwan, Associate professor, Chulalongkorn University
Other Study IDs: IRB No. 469/62
Record Dates: First submitted 2020-04-10; First posted 2020-04-17 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Ocular Surface Disease; Osteoarthritis; Diacerein
Keywords: Dry Eye Syndromes; Osteoarthritis; Ocular surface inflammation; Interleukin-1; Interleukin-1 receptor antagonist
MeSH Terms: conditions — Osteoarthritis; Dry Eye Syndromes | interventions — diacerein

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tears within Schirmer paper
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diacerein group: Osteoarthritis and dry eye patients treated with Diacerein
  Interventions: Drug: Diacerein

INTERVENTIONS:
Drug: Diacerein — Diacerein prescribing by orthopedist. Dry eye sign and symptom was asses before start diacerein and after 2 months.

SUMMARY:
Dry eyes is multi-factorial disease which inflammation play etiological role. Diacerein is drug which has anti-inflammatory effect by antagonist Interleukin-1, decrease Interleukin-1 receptor, increase Interleukin-1 Receptor antagonist. This observational study enrolled participants who going to take diacerein for osteoarthritis, measure corneal staining score, Ocular surface disease index score, Tear Osmolarity, Tear break up time, Schirmer 1 test, Interleukin-1 Receptor antagonist, Interleukin-1 alpha, Interleukin-1 beta level in tear at the time of enrollment and after 2 months.

ELIGIBILITY:
Inclusion Criteria:

1. Osteoarthritis with
2. Ocular surface index score ≥ 13 with
3. Corneal staining score ≥ 3

Exclusion Criteria:

1. Allergic to diacerein
2. Use Cyclosporin within 30 days
3. Eyelid problem
4. Change artificial tear while in the study
5. Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with osteoarthritis that prescribed Diacerein at out-patient clinic, Department of Orthopedic, King Chulalongkorn Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Corneal staining score change from baseline at 2 months | At the time of enrollment and 2 months
  Stain Cornea with Fluorescine, count and score staining at the cornea according to National eye institute : score 0-15 (0=no staining)

SECONDARY OUTCOMES:
Ocular surface disease index score | At the time of enrollment and 2 months
  Ocular Surface Disease Index : 0-100 (0=no any symptom)
Tear Osmolarity | At the time of enrollment and 2 months
  Use Tearlab to measure tear osmolarity
Tear break up time | At the time of enrollment and 2 months
  Stain Cornea with Fluorescine, wait until tear film break, record time that tear break
Schirmer 1 test | At the time of enrollment and 2 months
  place Schirmer strip at the fornix without anesthesia, wait for 5 min, record tear distance
Interleukin-1 receptor antagonist, Interleukin-1 alpha, Interleukin-1 beta level in tear | At the time of enrollment and 2 months
  Extract tear from Schirmer strip and use Bioplex for cytokine measurement of Interleukin-1 receptor antagonist(picogram/ml), Interleukin-1 alpha(picogram/ml), Interleukin-1 beta(picogram/ml)

CONTACTS AND LOCATIONS:
Overall Officials: Ngamjit Kasetsuwan, Principal Investigator — Department of Ophthalmology, Chulalongkorn University
Locations (1):
- Faculty of medicine, Chulalongkorn university, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided